CLINICAL TRIAL: NCT01486069
Title: Evaluation of the Perioperative Mandibular Positional Stability in Subjects With Dentofacial Deformity
Brief Title: Mandibular Stability and Dentofacial Deformity
Status: Completed | Type: Observational
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Alexandre Meireles Borba, Principal Investigator - PhD Student in Oral and Maxillofacial Surgery, University of Sao Paulo
Other Study IDs: FOUSP - PhD Surg - 01
Record Dates: First submitted 2011-12-02; First posted 2011-12-06 (Estimated); Last update posted 2013-06-14 (Estimated); Status verified 2013-06

CONDITIONS: Maxillofacial Abnormalities
Keywords: Dentofacial Deformity; Orthognathic Surgery; Mandible; Orthognathic Surgical Procedures
MeSH Terms: conditions — Maxillofacial Abnormalities; Dentofacial Deformities

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Dentofacial Deformity: Patients with dentofacial deformities candidate to orthognathic surgery

SUMMARY:
The present study intends to clarify whether there is positional mandibular stability in patients to be submitted to orthognathic surgery. In case of any instability exists, it is needed to understand if this could be related to a particular type of dentofacial deformity or could have any short-term or long-term influence on outcomes of the orthognathic surgery.

DETAILED DESCRIPTION:
Treatment of skeletal discrepancy nowadays is mainly performed by combination of clinical and surgical procedures in which orthodontics intends to align the teeth according to their respective alveolar bone and the surgical procedure - orthognathic surgery - realign the jaws in an adequate position among themselves and related to the rest of the craniofacial skeleton. Orthognathic surgery has developed throughout the years technically as well as regarding fixation devices for the operated segments, providing prediction of results with a low complication incidence. A debate point is related to the possible instability of the mandibular position as a reference for surgical planning due to its articulation with the temporal fossa, the temporomandibular joint. However, studies have shown that not always the mandible position obtained for the articulator reflects the position observed in subjects after induction of general anesthesia. Since there is no evidence that indicates that any alteration of the position of the mandible could influence the outcomes of a orthognathic surgery nor any relationship of a certain type of dentofacial deformity that would be beneficiated by an specific order of surgery or skeletal reference (maxilla or mandible), the present study intends to clarify some of these questions.

ELIGIBILITY:
Inclusion Criteria:

* Dentofacial Deformity candidate to orthognathic surgery;
* Systemically capable to be submitted to the orthognathic surgery.

Exclusion Criteria:

* Patient's health condition is not stable enough to guarantee uneventful outcome;
* Required data unable to be achieved;
* Patient not agreeing to participate to the study.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Data will be obtained from subjects to be submitted to orthognathic surgery by the Department of Oral & Maxillofacial Surgery of the Hospital Geral Universitário of the city of Cuiabá - Brazil during the period of March 2012 through March 2013. Considering the local demand, thirty subjects are expected to be included in the research.
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2012-07; Primary Completion 2013-02 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Variability in mandibular position for different dental occlusion registrations | Perioperative to orthognathic surgery
  Centric occlusion, maximum intercuspation and occlusion under general anesthesia

CONTACTS AND LOCATIONS:
Overall Officials: Alexandre M Borba, DDS, MSc, Principal Investigator — University of Sao Paulo
Locations (1):
- Hospital Geral Universitario, Cuiabá, Mato Grosso, Brazil

REFERENCES:
- [Background] Bamber MA, Abang Z, Ng WF, Harris M, Linney A. The effect of posture and anesthesia on the occlusal relationship in orthognathic surgery. J Oral Maxillofac Surg. 1999 Oct;57(10):1164-72; discussion 1172-4. doi: 10.1016/s0278-2391(99)90476-7. PMID 10513861
- [Background] Posnick JC, Ricalde P, Ng P. A modified approach to "model planning" in orthognathic surgery for patients without a reliable centric relation. J Oral Maxillofac Surg. 2006 Feb;64(2):347-56. doi: 10.1016/j.joms.2005.10.022. No abstract available. PMID 16413911
- [Background] Turvey T. Sequencing of two-jaw surgery: the case for operating on the maxilla first. J Oral Maxillofac Surg. 2011 Aug;69(8):2225. doi: 10.1016/j.joms.2010.10.050. Epub 2011 Feb 3. No abstract available. PMID 21295393
- [Background] Perez D, Ellis E 3rd. Sequencing bimaxillary surgery: mandible first. J Oral Maxillofac Surg. 2011 Aug;69(8):2217-24. doi: 10.1016/j.joms.2010.10.053. Epub 2011 Feb 3. No abstract available. PMID 21292376
- [Background] Weffort SY, de Fantini SM. Condylar displacement between centric relation and maximum intercuspation in symptomatic and asymptomatic individuals. Angle Orthod. 2010 Sep;80(5):835-42. doi: 10.2319/090909-510.1. PMID 20578853